CLINICAL TRIAL: NCT03784898
Title: Collection of Blood Samples From Patients With Relapsing Forms of Multiple Sclerosis (RMS) Who Have Developed Immune Thrombocytopenic Purpura (ITP) After LEMTRADA® Treatment
Brief Title: Collection of Blood Samples From Patients With Relapsing MS Who Developed ITP After Receiving Lemtrada
Acronym: LEMTRADA-ITP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASY15905; U1111-1225-1333
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants Diagnosed With ITP (Other): Participants with RMS who developed ITP after Lemtrada treatment were included in this study and provided blood samples for future genetic testing and biomarker analysis.
  Interventions: Other: Blood draw for future biomarker analysis

INTERVENTIONS:
Other: Blood draw for future biomarker analysis — Each participant was required to undergo blood draw for future genetic testing and biomarker analysis as mentioned in the informed consent form (ICF).

SUMMARY:
Primary Objective:

To collect blood samples in a new cohort of Relapsing Forms of Multiple Sclerosis (RMS) participants who had developed immune thrombocytopenic purpura (ITP) after LEMTRADA treatment, for future Deoxyribonucleic acid (DNA) analysis as part of a global biomarker project assessing pre-identified candidate single nucleotide polymorphisms (SNPs) associated to the development of ITP after LEMTRADA treatment in RMS participants.

DETAILED DESCRIPTION:
One to 70 days, as screening and inclusion visit(s) were performed the same day or on separate days with a maximum timeframe of 30 days apart. One visit was required for blood draw. However, if a second visit occured, it took place within 40 days of the first visit.

ELIGIBILITY:
Inclusion criteria :

* Male and female adult participants who had been treated with LEMTRADA, with development of ITP subsequent to treatment. Participants does not need to be currently on LEMTRADA treatment.
* Participants who had signed the study ICF.

Exclusion criteria:

- Not applicable

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 8400001, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single site in the United States. A total of 14 participants were screened between 8 February 2019 to 11 December 2019, of which,1 participant was screen failure. Screen failures was mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 13 participants were enrolled in the study.
Groups:
- Participants Diagnosed With ITP: Participants with Relapsing Forms of Multiple Sclerosis (RMS) who developed Immune thrombocytopenic purpura (ITP) after Lemtrada treatment were included in this study and provided blood samples for future genetic testing and biomarker analysis.
Period: Overall Study
Arm/Group | Participants Diagnosed With ITP
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | Participants Diagnosed With ITP
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Provided Whole Blood Samples for DNA Extraction and Analysis
Description: Each participant provided a maximum total of 69 milliliter of whole blood sample. Samples were collected in the following order: 1. Deoxyribonucleic acid (DNA) Paired box (PAX)gene tubes (2 tubes), 2. Ribonucleic acid (RNA) PAXgene tubes (2 tubes), 3. Ethylenediaminetetraacetic acid (EDTA) tubes for peripheral blood mononuclear cells (PBMCs) (5 tubes), 4. Serum Separator tube (SST) (1 tube), and 5. Dipotassium Ethylenediaminetetraacetic acid (K2EDTA) tube (1 tube); where DNA PAXgene tubes were used for DNA preparation, RNA PAXgene tubes for RNA preparation, EDTA for PBMC isolation, SST tubes for serum preparation and K2EDTA for plasma preparation. DNA was extracted from peripheral blood for future analysis.
Time Frame: Baseline (Day 1)
Population: Analysis was performed on all enrolled population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Diagnosed With ITP
Number analyzed (Participants) | 13
Participants
  DNA PAXgene (tube 1) | 12
  DNA PAXgene (tube 2) | 12
  RNA PAXgene (tube 1) | 12
  RNA PAXgene (tube 2) | 12
  EDTA for PBMCs (tube 1) | 13
  EDTA for PBMCs (tube 2) | 13
  EDTA for PBMCs (tube 3) | 13
  EDTA for PBMCs (tube 4) | 13
  EDTA for PBMCs (tube 5) | 5
  SST tube | 12
  K2EDTA tube | 12

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from the signature of the Informed consent form until the end of the study (i.e. up to 307 days)
Description: Analysis was performed on all enrolled participants.
Arm/Group | Participants Diagnosed With ITP
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03784898/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03784898/SAP_001.pdf